CLINICAL TRIAL: NCT00842153
Title: A Study to Evaluate the Efficacy and Tolerability of Clobetasol Propionate vs. Vehicle in the Treatment of Mild to Moderate Plaque-Type Psoriasis
Brief Title: Evaluation of the Efficacy and Tolerability of Clobetasol Propionate Foam Compared to Vehicle Foam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OEF0701
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Type Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clobetasol Propionate Foam (Experimental): Topical foam formulation that includes clobetasol propionate (Steroid)
  Interventions: Drug: Clobetasol propionate foam
- Vehicle Foam (Placebo Comparator): Vehicle foam is the same as the clobetasol propionate foam except it does not include the active drug.
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Clobetasol propionate foam — Topical Clobetasol propionate foam
  Other Names: Olux-E
  Arms: Clobetasol Propionate Foam
Drug: Vehicle foam — Vehicle foam does not include the active drug.
  Arms: Vehicle Foam

SUMMARY:
The purpose of the study is to compare the efficacy and safety of Clobetasol propionate to that of its Vehicle in the treatment of mild to moderate plaque-type psoriasis.

DETAILED DESCRIPTION:
The purpose of the study is to compare the efficacy and safety of Clobetasol propionate to that of its Vehicle in the treatment of mild to moderate plaque-type psoriasis. This is a multi-center, double blind, randomized, parallel designed study which consists of 2 weeks of treatment and a follow-up visit 2 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, and at least 12 years of age. Female subjects of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study.
* Mild to moderate, plaque-type psoriasis
* Target lesion on the trunk or extremities (excluding palms/soles, elbows, or knees) with a score of 2 or 3 for each of erythema, scaling and plaque thickness
* Able to understand the requirements of the study and sign Informed Consent/HIPAA Authorization Forms. Subjects under the legal age of consent in the state where the study is conducted must also have the written, informed consent of a parent or legal guardian.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test) breast feeding or who are of childbearing potential and not practicing a reliable method of birth control
* Known allergy to clobetasol propionate or other topical corticosteroids; or to any component of the investigational formulations
* Subjects who have not complied with the proper wash-out periods for prohibited medications
* Medical condition that in the opinion of the investigator, contraindicates the subject's participation in the clinical study
* Skin disease/disorder that might interfere with the study related diagnosis or evaluations
* Evidence of recent alcohol or drug abuse
* History of poor cooperation, non-compliance with medical treatment or unreliability

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Center for Dermatology, Cosmetic and Laser, Fremont, California
  - Dermatology Specialists, Louisville, Kentucky

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A wash-out period of 2 to 8 weeks, the duration of which varied by specific medication, was required prior to Visit 1.
Groups:
- Olux-E Foam: Olux-E foam containing 0.05% clobetasol propionate, applied twice daily (morning and evening [BD]) for four weeks to the affected area on the scalp and body
- Vehicle Foam: Vehicle foam without the active ingredient clobestasol propionate, applied BD for four weeks to the affected area on the scalp and body
Period: Overall Study
Arm/Group | Olux-E Foam | Vehicle Foam
Started | 28 | 30
Completed | 27 | 27
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olux-E Foam | Vehicle Foam | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (20.0) | 47.2 (13.4) | 50.6 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 23 | 46
  Black | 1 | 0 | 1
  Hispanic | 0 | 2 | 2
  Asian | 2 | 3 | 5
  Other (not included above; including mixed race) | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Target Lesion Global Improvement (TLGI) Score of 0, 1, or 2 at Weeks 1, 2, and 4
Description: The investigator assessed the TLGI of participants relative to their initial Baseline condition based on a 7-point scale: 0=completely cleared, possible residual discoloration; 1=almost cleared, 90% improvement, very significant clearance with only traces of disease remaining; 2=marked improvement, approximately 75%, with some disease remaining; 3=moderate improvement, approximately 50%; 4=mild improvement, approximately 25%, significant disease remains; 5=no change, no detectable improvement; 6=excerbation, worsening of signs and symptoms of disease.
Time Frame: Weeks 1, 2, and 4
Population: Intent-to-Treat (ITT) Population: all enrolled participants. Participants who returned for the visit specified (Week 1, 2, and/or 4) were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 27 | 30
participants
  Week 1, n=26, 30 | 6 | 2
  Week 2, n=26, 30 | 19 | 3
  Week 4, n=27, 28 | 12 | 2
Statistical Analysis 1: Comparison: Olux-E Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.1269, Fisher Exact — P-value for Week 1
Statistical Analysis 2: Comparison: Olux-E Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.0001, Chi-squared — P-value for Week 2
Statistical Analysis 3: Comparison: Olux-E Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.0015, Chi-squared — P-value for Week 4

2. Secondary Outcome: Number of Participants With a TLGI Score of 0, 1, 2, or 3 at Weeks 1, 2, and 4
Description: as for outcome 1
Time Frame: Weeks 1, 2, and 4
Population: ITT Population. Participants who returned for the visit specified (Week 1, 2, and/or 4) were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 27 | 30
participants
  Week 1, n=26, 30 | 19 | 6
  Week 2, n=26, 30 | 21 | 9
  Week 4, n=27, 28 | 15 | 8

3. Secondary Outcome: Number of Participants With a Pruritus (Overall) Score of 0 or 1 at Week 2
Description: Participants assessed their level of pruritus (itching) over the previous 24-hour period using the following scale: 0=no itching; 1=minimal, very rarely aware of localized itching, present when relaxing and lasted for very short time; 2=mild, aware of itching at times, present when relaxing, not present when focused on other activities; 3=moderate, often aware of itching, annoying, sometimes disturbed sleep and daytime activities; and 4=severe, constant itching, distressing, frequent sleep disturbance, interfered with activities.
Time Frame: Week 2
Population: ITT Population. Participants who returned for the visit specified (Week 2) were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 30
participants | 21 | 17

4. Secondary Outcome: Number of Participants With an Erythema Score of 0 or 1 at Week 2
Description: The investigator individually graded the severity of erythema (redness of skin) in participants as: 0=hyperpigmentation, pigmented macules (flat, distinct, colored area of skin), diffuse faint pink or red coloration; 1=no evidence of erythema, hyperpigmentation present; 2=faint erythema; 3=light red coloration; 4=moderate red coloration; and 5=bright red coloration.
Time Frame: Week 2
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 30
participants | 6 | 1

5. Secondary Outcome: Number of Participants With a Scaling Score of 0 or 1 at Week 2
Description: The investigator individually graded the severity of scaling in participants as: 0=no scaling; 1=no evidence of scaling; 2=minimal, occasional fine scale over less than 5% of the lesion; 3=mild, fine scales predominate; 4=moderate, coarse scales predominate; and 5=marked, thick nontenacious scales predominate.
Time Frame: Week 2
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 30
participants | 11 | 5

6. Secondary Outcome: Number of Participants With a Plaque Thickness Score of 0 or 1 at Week 2
Description: The investigator individually graded the severity of plaque thickness in participants as: 0=no elevation over normal skin; 1=possible but difficult to ascertain whether there is a slight elevation above normal skin; 2=slight but definite elevation, typically edges are indistinct or sloped; 3=moderate elevation with rough or sloped edges; 4=marked elevation typically with hard or sharp edges; and 5=very marked elevation typically with hard, sharp edges.
Time Frame: Week 2
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 30
participants | 16 | 4

7. Secondary Outcome: Number of Participants With a Score of 0 or 1 for Subject Global Assessment at Week 2
Description: Participants assessed all treated areas using the Subject Global Assessment scale: 0=skin completely clear, possible residual hyperpigmentation; 1=psoriasis almost clear, patchy remnants of fine scaling present; 2=psoriasis mild, with small amount of psoriasis remaining (i.e., fine to coarse scales in some areas, definite redness, barely visible plaque thickness); 3=psoriasis moderate, between slight and definitely noticeable; 4=psoriasis very noticeable with redness, scaling, plaque thickness; 5=psoriasis severe with severe redness, thick scaling, and plaques.
Time Frame: Week 2
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 30
participants | 5 | 1

8. Secondary Outcome: Mean Percent Change From Baseline to Week 2 in Pruritus (Target Lesion)
Description: Participants assessed their level of pruritus (itching) for the target lesion using a 10 centimeter (cm) Visual Analogue Scale (VAS) with the left side anchored with "0=None" and the right side anchored with "10=Very Severe." A target lesion (>2 cm squared [cm^2]) was considered to be one on the trunk or extremities (excluding palms/soles, elbows, or knees). Percent change from Baseline was calculated as the value at Week 2 minus the value at Baseline (Week 0) divided by the Baseline (Week 0) value * 100.
Time Frame: Baseline (Week 0) and Week 2
Population: ITT Population. Participants who returned for the visit specified (Week 2) and/or provided an assessment of pruritis were evaluated; not all participants returned for every study visit.
Measure: Mean (Standard Deviation); unit: Percent change in scores on a scale
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 25 | 25
Percent change in scores on a scale | -30.5 (155.8) | 40.1 (442.0)

9. Secondary Outcome: Mean Percent Change From Baseline to Week 2 in Percent (%) of Body Surface Area (BSA) Affected
Description: Percent change from Baseline was calculated as the value at Week 2 minus the value at Baseline (Week 0) divided by the Baseline (Week 0) value * 100. Data for this outcome measure were not collected; thus, no data were analyzed.
Time Frame: Baseline (Week 0) and Week 2
Population: ITT Population
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With a TLGI Score of 0, 1, or 2 at Week 1 and Week 4
Description: as for outcome 1
Time Frame: Week 1 and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 1 and/or 4) and/or provided an assessment for pruritus were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 27 | 30
participants
  Week 1, n=26, 30 | 6 | 2
  Week 4, n=27, 28 | 12 | 2

11. Secondary Outcome: Number of Participants With a Pruritus (Overall) Score of 0 or 1 at Baseline and Week 4
Description: as for outcome 3
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population Participants who returned for the visit specified (Week 4) and/or provided an assessment for pruritus were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 28 | 30
participants
  Baseline (Week 0), n=28, 30 | 8 | 9
  Week 4, n=27, 28 | 19 | 17

12. Secondary Outcome: Number of Participants With an Erythema Score of 0 or 1 at Baseline and Week 4
Description: as for outcome 4
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 4) and/or provided an assessment for erythema were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 28 | 30
participants
  Baseline (Week 0), n=28, 30 | 0 | 0
  Week 4, n=27, 28 | 6 | 1

13. Secondary Outcome: Number of Participants With a Scaling Score of 0 or 1 at Baseline and Week 4
Description: as for outcome 5
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 4) and/or provided an assessment for scaling were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 28 | 30
participants
  Baseline (Week 0), n=28, 30 | 0 | 0
  Week 4, n=27, 28 | 6 | 4

14. Secondary Outcome: Number of Participants With a Plaque Thickness Score of 0 or 1 at Baseline and Week 4
Description: as for outcome 6
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 4) and/or provided an assessment for plaque thickness were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 28 | 30
participants
  Baseline (Week 0), n=28, 30 | 0 | 0
  Week 4, n=27, 28 | 12 | 2

15. Secondary Outcome: Number of Participants With a Score of 0 or 1 for Subject Global Assessment at Baseline and Week 4
Description: as for outcome 7
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 4) and/or provided an assessment for Subject Global Assessment were evaluated; not all participants returned for every study visit.
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 28 | 30
participants
  Baseline (Week 0), n=28, 30 | 0 | 0
  Week 4, n=27, 28 | 7 | 1

16. Secondary Outcome: Mean Percent Change From Baseline to Week 4 in Pruritus (Target Lesion)
Description: Participants assessed their level of pruritus (itching) for the target lesion using a 10 centimeter (cm) Visual Analogue Scale (VAS) with the left side anchored with "0=None" and the right side anchored with "10=Very Severe." A target lesion (>2 cm squared [cm^2]) was considered to be one on the trunk or extremities (excluding palms/soles, elbows, or knees). Percent change from Baseline was calculated as the value at Week 4 minus the value at Baseline (Week 0) divided by the Baseline (Week 0) value * 100.
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population. Participants who returned for the visit specified (Week 4) and/or provided an assessment for pruritus were evaluated; not all participants returned for every study visit.
Measure: Mean (Standard Deviation); unit: Percent change in scores on a scale
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 26 | 23
Percent change in scores on a scale | -6.8 (213.5) | -40.2 (67.4)

17. Secondary Outcome: Mean Percent Change From Baseline to Week 4 in Percent (%) of Body Surface Area (BSA) Affected
Description: Percent change from Baseline was calculated as the value at Week 4 minus the value at Baseline (Week 0) divided by the Baseline (Week 0) value * 100. Data for this outcome measure were not collected; thus, no data were analyzed.
Time Frame: Baseline (Week 0) and Week 4
Population: ITT Population
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: One participant in the ITT Population was dispensed study drug but did not return after the Baseline visit; thus, this participant was not included in the analysis of serious adverse events (SAEs) or non-serious AEs.
Arm/Group | Olux-E Foam | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 3/27 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olux-E Foam (N=27) | Vehicle Foam (N=30)
Tooth Extraction Surgery (General disorders) | 1 | 0
Common Cold (Infections and infestations) | 1 | 0
Hemorrhoids (General disorders) | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Diagnosed Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Moderately Elevated Prostate-Specific Antigen (PSA) (General disorders) | 0 | 1
Worsening Of Psoriasis, Upper Extremities (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrointestinal Virus (Infections and infestations) | 0 | 1
Papular Dermatitis On Left Upper Abdomen (Skin and subcutaneous tissue disorders) | 0 | 1
Left Shin, Target Area Worse, Severe Itching/Oozing/Wheeping (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.